CLINICAL TRIAL: NCT03680937
Title: Methods for Fertility Preservation: Impact of Vitrification on in Vitro Matured Oocytes
Acronym: OVOMIV
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: CHU-393
Record Dates: First submitted 2018-06-05; First posted 2018-09-21 (Actual); Last update posted 2018-09-21 (Actual); Status verified 2018-09

CONDITIONS: Fertility; Cancer
Keywords: Vitrification; In vitro maturation; time lapse; High resolution imaging; quantitative molecular analysis
MeSH Terms: conditions — Neoplasms | interventions — Vitrification

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Immature oocytes vitrified before in vitro maturation: Immature oocytes will be vitrified using closed system vitrification with a semiautomatic method. After warming, a maturation culture will be performed during 36 hours
  Interventions: Other: Gavi , Merck® (automated vitrification instrument); Other: Vitrification
- Immature oocytes vitrified after in vitro maturation: A maturation culture of immature oocytes will be performed in vitro during 36 hours. After IVM, mature oocytes will be vitrify in closed system by a semi-automatic method.
  Interventions: Other: Gavi , Merck® (automated vitrification instrument); Other: Vitrification
- Fresh oocytes: The culture of immature oocytes will be performed during 36 hours

INTERVENTIONS:
Other: Gavi , Merck® (automated vitrification instrument) — Gavi, Merck ® permits semi-automated vitrification with closed system.
  Groups: Immature oocytes vitrified after in vitro maturation; Immature oocytes vitrified before in vitro maturation
Other: Vitrification — Group 1: immature ovocytes vitrified before IVM; Group 2: immature oocytes vitrified after IVM; Group3: fresh immature oocytes treated by IVM (without vitrification, control group).
  Groups: Immature oocytes vitrified after in vitro maturation; Immature oocytes vitrified before in vitro maturation

SUMMARY:
During the last decades, there was an improvement of the cancer treatments of the woman and the teenagers. Therefore higher survival rate is described. However, cancer treatments can alter the reproduction functions and reduce considerably the window of the fertility to the adulthood. Therefore, it is recommended to proceed to a fertility preservation by oocytes vitrification when it is possible. The vitrification is a freezing technique allowing high survival rate and similar results by assisted reproductive technologies compared with the use of fresh oocytes. An innovative method of automated vitrification was recently developed. The usual protocol consist to vitrify mature oocytes. However, this strategy cannot be used for hormone -sensitive cancer or when ovarian stimulation is not possible. In these situations, immature oocytes can be collected. It is also necessary to realize an in vitro maturation step for a use by assisted reproductive technology.

According to the recent data of the literature, it remains unclear whether the vitrification of ovocytes must be performed before or after in vitro maturation (IVM). Therefore the aim of this study is to study the impact on structure and functions of ovocytes when vitrification is performed before or after IVM. The vitrification will be performed by a semi-automatic method which is an innovative method.

DETAILED DESCRIPTION:
To perform this study, investigator will compare three groups. Group 1: immature ovocytes vitrified before IVM; Group 2: immature oocytes vitrified after IVM; Group3: fresh immature oocytes treated by IVM (without vitrification, control group).

The immature oocytes provide from ICSI patients. In routine these oocytes (germinal vesicle) are normally destroyed because they cannot be used for injection. The women will give an informed and written consent. Inclusion criteria are women less 37 years without dysovulation.

The vitrification will be performed with the semi-automatic method (Gavi, Merck). The kinetic and maturation rate will be analysed by time lapse (Primovision, Vitrolife) In the mature oocytes, the actin and tubulin cytoskeleton, the spindle organization and the cortical granules will be studied by immunofluorescence and 3D confocal microscopy. The expression of maternal factors transcription will be analyzed by RT-PCR. The ploidy will be analysed by multiFISH and/or CGH array.

ELIGIBILITY:
Inclusion Criteria:

* ICSI treatment
* Immature oocytes
* Without ovulation pathologies

Exclusion Criteria:

* Polykistic ovarian syndrome
* Endometriosis
* Ovulatory disease

Ages: 18 Years to 37 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: women
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2018-09-20 (Estimated); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-07-31 (Estimated)

PRIMARY OUTCOMES:
The embryonic development kinetics | 6 days after ICSI and through study completion
  from the records obtained with Time Lapse Primovision, investigator will be able to determine the precise times of embryonic development after in vitro maturation.

SECONDARY OUTCOMES:
Analysis of actin and tubulin cytoskeleton and spindle organization in mature ovocytes (Metaphase II) | 01/01/2019 - 31/12/2019
  Metaphase-II stage oocytes will be used for Immuno-Fluorescence experiments to stain actin, tubulin and chromosomes. Oocytes will be imaged using confocal microscope to perform high resolution imaging and quantitative image analysis. The length, position and orientation of the second meiotic spindle will be analysed. The actin network and chromosomes will be analysed quantitatively. All measurements will be compared with fresh matured (Metaphase-II) oocytes used as a control group.
Analysis of chromosome segregation during the first meiotic division | 01/01/2019 - 31/12/2019
  A multi Fluorescence in Situ Hybridization and/or a CGH array will be performed to measure the chromosome segregation after vitrification
Analysis of cortical granules distribution in mature (Metaphase II) oocytes. | 01/01/2019 - 31/12/2019
  A staining with Lectin will be used to mark cortical granules of matured oocytes to observe whether the protocol has an impact on their spatial distribution. To analyse this staining, investigator will use quantitative image analysis method.
Analysis of maternal factor stabilities. | 01/01/2019 - 31/12/2019
  Maternal factors stored in the oocyte cytoplasm during oogenesis as proteins and transcripts are essential for the early embryonic development. Investigator will perform Reverse Transcription combined with Real Time PCR to quantify transcript amounts of candidates genes selected from human oocytes databases.

CONTACTS AND LOCATIONS:
Overall Officials: Florence BRUGNON, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- Chu Clermont-Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Derived] Chaput L, Dollet S, Eymard-Pierre E, Pereira B, Lucas C, Gremeau AS, Tchirkov A, Marteil G, Brugnon F. Analysis of maturation dynamics and oocyte nuclear quality after rescue-IVM and semi-automated vitrification. Hum Reprod. 2025 Jul 1;40(7):1344-1356. doi: 10.1093/humrep/deaf078. PMID 40373183